CLINICAL TRIAL: NCT05796843
Title: 360 Degrees Virtual Reality-based Mirror Therapy for Upper Extremity Rehabilitation Among Stroke Patients
Brief Title: 360 Degrees Virtual Reality-based Mirror Therapy for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Sungbae Jo, Physical Therapist, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYU 2023-01-009-001
Record Dates: First submitted 2023-03-16; First posted 2023-04-04 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Stroke Rehabilitation; Mirror Movement Therapy
Keywords: Stroke; Stroke Rehabilitation; Mirror Movement Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 360 Degrees Virtual Reality-based Mirror Therapy Group (Experimental): The group which will receive 360 Degrees Virtual Reality-based Mirror Therapy Group
  Interventions: Procedure: 360 Degrees virtual reality-based mirror therapy; Procedure: Conventional Physical Therapy
- Traditional Mirror Therapy Group (Active Comparator): The group which will receive traditional mirror therapy using a conventional mirror
  Interventions: Procedure: Traditional mirror therapy; Procedure: Conventional Physical Therapy
- Conventional Physical Therapy Group (Active Comparator): The group which will receive conventional rehabilitation for upper extremity
  Interventions: Procedure: Conventional Physical Therapy

INTERVENTIONS:
Procedure: 360 Degrees virtual reality-based mirror therapy — Participants will receive mirror therapy using a virtual reality device (Pico G2 VR 4K, Pico, China). They will be asked to follow tasks that are played in HMD using their paralyzed hand. The video played using HMD will be video taped using 360 degree camera prior to the treatment. The 360MT will last 30 minutes/session, 3 sessions a week for 4 weeks. The tasks are finger flexion-extension, wrist flexion-extension and pronation-supination, and elbow flexion-extension for ten repetitions.
  Arms: 360 Degrees Virtual Reality-based Mirror Therapy Group
Procedure: Traditional mirror therapy — Participants will receive mirror therapy using an acrylic mirror (40cm x 40cm x 3cm) that reflects unparalyzed side of them. They will be asked to perform tasks including finger flexion-extension, wrist flexion-extension and pronation-supination, and elbow flexion-extension for ten repetitions. They will be asked to follow the reflection on mirror using their paralyzed limb. The TMT will last 30 minutes/session, 3 sessions a week for 4 weeks.
  Arms: Traditional Mirror Therapy Group
Procedure: Conventional Physical Therapy — Participants will receive conventional physical therapy including neurodevelopmental therapy, muscle strengthening exercises, and joint mobilization which will be provided 60 minutes per day, 5 sessions a week, for 4 weeks. The therapy will follow upper extremity rehabilitation protocol which consists of three phases of warm up, circuit, and cool down exercises

SUMMARY:
The goal of this randomized controlled trial is to compare the effects of 360 degree virtual reality-based mirror therapy (360MT) to traditional mirror therapy (TMT) and conventional physical therapy (control group) on upper extremity function among stroke patients.

The main questions it aims to answer are:

* Would 360MT be more effective when treated for 4 weeks in outcome measure ments including: Fugl-Meyer Assessment for upper extremity (FMA-UE); manual function test (MFT); and box & block test (BBT)?
* How would particants' experience be in terms of satisfactory and enjoyment during 360MT?

The study will have three groups of participants who will be involved in different tasks:

* 360MT group: will receive mirror therapy using a virtual reality device (HMD) and perform tasks with their paralyzed hand. Sessions will last 30 minutes, 3 times a week for 4 weeks.
* TMT group: will receive mirror therapy using an acrylic mirror and perform finger, wrist, elbow exercises using their paralyzed limb. Sessions will last 30 minutes, 3 times a week for 4 weeks.
* Control group: will receive conventional physical therapy consisting of exercises for the upper extremity, 60 minutes per day, 5 sessions a week, for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* who have not passed 12 months since onset;
* who can understand and follow instructions;
* who have ≥21 scores in Korean version of Mini-Mental State Examination (MMSE-K);
* who have mild to moderate motor impairment according to the Fugl Meyer Assessment (FMA) scores

Exclusion Criteria:

* patients who have any kinds of mental disorder and/or Alzheimer's disease;
* who have orthopedic and/or musculoskeletal injury;
* who have apraxia; and
* who have previous experiences of participating in investigations and/or mirror therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for upper extremity (FMA-UE) | Changes from baseline after 4 weeks of intervention
  The test is one of the most frequently used evaluation tools that quantitatively assesses recovery after stroke by measuring motor skills, balance ability, sensory function, and range of motion. The maximum total score for FMA-UE is 66 points, containing 18 items to evaluate shoulder, elbow, and forearm; 5 for the wrist; 7 for the hand; and 3 items for coordination.

SECONDARY OUTCOMES:
Manual Function Test (MFT) | Changes from baseline after 4 weeks of intervention
  This test can reflect the degree of upper extremity dysfunction after stroke, consists of four items each for shoulder and hands. The MFT has a maximum total score of 32 points
Box & Block Test (BBT) | Changes from baseline after 4 weeks of intervention
  used to evaluate manual dexterity of the hands. The evaluation involves wooden blocks (2.5 cm3) placed in a box (53.7cm x 8.5 cm x 27.4cm) which is divided by a partition in the center. The subjects were instructed to move as many boxes as possible from one side to another in one minute using their affected upper limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Sungbae Jo, PhD candidate, Principal Investigator — Sahmyook University
Locations (1):
- Myeonji Choonhae Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No